CLINICAL TRIAL: NCT05614609
Title: Discomfort in Upper Airways Due to intubation-a Randomized Controlled Trial in a Norwegian Hospital
Brief Title: Discomfort in Upper Airways Due to intubation-a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold University College (Other)
Responsible Party: Principal Investigator, Ann-Chatrin Leonardsen, Professor, Ostfold Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Sykehuset Østfold
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Complications; Intubation; Difficult or Failed; Intubation Complication
MeSH Terms: conditions — Postoperative Complications | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Block randomization through randomization.com. Proprotion of hoarseness grade-2-or-3 = 30 % in spray and 10 % in rocuronium.
  59 patients in each arm.
  "sig p <= ,05", H0 = 0 + 1,96*√[30(100-30)n + 10(100-10)/n] Gitt "power >= ,80" , HAlt = (30-10) - 0,84*√[30(100-30/n) + 10(100- 10/n)]
Who Masked: Participant, Care Provider
Masking Description: A study nurse will prepare sealed envelopes with the study-arm specified inside. Patients fullfilling the inclusion criteria will be invited to participate. Patients will be blinded for study arm. Intubation will be performed by trained intubators. However, due to the medications possible risk for rest-curarisation, the anesthesia personnel will possibly be able to detect intervention. However, care personnel collecting data will not know which study arm the patient belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine spray on the glottis (Active Comparator): Lidocaine 20 mgl/ml- 4,4 ml will be sprayed on the glottis. Ventilation for 90 sek, intubation
  Interventions: Drug: Lidocaine topical
- Muscle relaxing medication (Active Comparator): Rocuronium 0,6 mg/kg administered intravenous. Ventilation for 2.5 minutes (150seconds), intubation
  Interventions: Drug: Lidocaine topical

INTERVENTIONS:
Drug: Lidocaine topical — Comparing lidocaine spray and muscle relaxing medication
  Other Names: Rocurinoum 0.6 mg/kg intravenous

SUMMARY:
Few studies have compared different methods for optimalizing intubation conditions in general anesthesia. This randomized controlled trial will compare two different methods for intubation in general anesthesia in gastro- or gynecological procedures.

DETAILED DESCRIPTION:
In general anesthesia, it is neccessary to secure the airways with an endotracheal tube. There is no international consensus on how intubation is most efficiently conducted. A cochrane review compared using muscular relaxing medication versus not using blocks for intubation. Primary outcomes were intubation conditions and discomfort in upper airways. The authors concluded that research is limited, and that further research is needed. No studies have compared local anesthetic spray on the glottis and muscular relaxing medication in intubation, focusing on discomfort in upper airways. The null-hypothesis of this study is that there is no difference in upper airway discomfort when using local anesthetic spray or muscular relaxing medication. The study will have a randomized controlled design, randomizing patients undergoing gastro- or gynecological procedures in general anesthesia to receiving either rocuronium (muscle relaxing medication) intravenous, or lidocain spray on the glottis before intubation. The primary outcome is postoperativ hoarseness one hour after intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Association of Anesthesiologists Classification system for physical status) I-III
* Understand and can express themselves in Norwegian
* Able to give informed consent to participate

Exclusion Criteria:

* Cave lidocain and/or muscle relaxing medication
* BMI above 40
* Anticipated difficult intubation
* Need for ventricular tube
* Pathology or malformations in upper airways

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Degree of hoarseness 1 hour after extubation | 1 hours
  Scored on a scale : 0=no, 1= self reported hoarseness, 2=observed hoarsness by care personnel, 3=aphonia

SECONDARY OUTCOMES:
Intubation conditions | Before intubation
  Cormack & Lehane four degrees
Number of intubation attempts | At intubation
  Number
Number of patients needing extra equipment for intubating | At intubation
  bourgie, c-mac, other
Proportion of patients who cough when spraying | At intubation
  yes/no
Proportion of patients with normal anatomy in upper airways | At intubation
  yes/no
Blood pressure changes during intubation | at intubation
  Blood pressure before and 2 minutes after intubation
Heart rate changes during intubation | at intubation
  Heart rate before and 2 minutes after intubation
Proportion of patients who cough on tube at extubation | At extubation
  yes/no
Proportion of patients with blood on tube after extubation | At extubation
  yes/no
Degree of hoarsness 24 and 48 hours after extubation | 2-48 hours
  Scored on a scale : 0=no, 1= self reported hoarseness, 2=observed hoarsness by care personnel, 3=aphonia
Proportion of patients reporting different degrees of sore throat at 2, 24 and 48 hours after extubation | 2-48 hours
  0=no, 1=mild, 2=moderate, constant pain when swallowing, 3=severe pain needing analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Ann-Chatrin Linqvist Leonardsen, Kråkerøy, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fjaerestad T, Oyras P, Solbakk KI, Leonardsen AL. Upper airway discomfort: a randomized controlled double-blind trial comparing rocuronium and lidocaine spray for intubation. Eur J Med Res. 2025 Jun 20;30(1):498. doi: 10.1186/s40001-025-02798-8. PMID 40542414